CLINICAL TRIAL: NCT01037959
Title: Randomized, Double-Blind, Placebo-Controlled Trial Assessing Norfloxacin in the Prevention of Complications in Patients With Cirrhosis and Severe Liver Failure
Brief Title: Norfloxacin Therapy for Patients With Cirrhosis and Severe Liver Failure
Acronym: NORFLOCIR
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: lack of recruitement
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: P071220
Record Dates: First submitted 2009-12-21; First posted 2009-12-23 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-11

CONDITIONS: Cirrhosis
Keywords: severe cirrhosis; Patients with severe cirrhosis
MeSH Terms: conditions — Fibrosis | interventions — Norfloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Norfloxacin (Active Comparator): Patients with severe cirrhosis treated with norfloxacin
  Interventions: Drug: Norfloxacin
- Placebo (Placebo Comparator): Patients with severe cirrhosis treated with placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Norfloxacin — 400 mg/day (per os) for 6 months
  Arms: Norfloxacin
Drug: Placebo — 1 pill/day (per os) for 6 months
  Arms: Placebo

SUMMARY:
Patients with advanced cirrhosis have abnormal translocation of Gram-negative bacteria across the intestinal barrier and subsequent systemic inflammatory response. We hypothesized that this translocation may worsen the underlying liver disease. Thus, the aim of this trial was to assess the effects of the oral administration of norfloxacin (an antibiotic that suppresses intestinal Gram-negative bacteria) on the development of complications of cirrhosis.

DETAILED DESCRIPTION:
Intestinal translocation of Gram-negative bacteria occurs in patients with advanced cirrhosis. Long-term oral administration of 400 mg/day of norfloxacin (a fluoroquinolone antibiotic) is known to induce selective intestinal decontamination against Gram-negative bacteria. A randomized, double-blind, placebo-controlled trial of oral norfloxacin (400 mg/day for 1 year) has been conducted in a small series of patients with advanced cirrhosis and low ascitic fluid protein concentrations <1.5 g/dL. This trial showed that norfloxacin therapy significantly increased the 1-year probability of being free of a first episode of spontaneous bacterial peritonitis (SBP) and improved 3-month survival. In this previous study, oral norfloxacin therapy was also found to decrease the risk of development of hepatorenal syndrome, a very severe complication of cirrhosis. It has been suggested that bacterial translocation, through the release of bacterial byproducts, results in systemic inflammation and subsequent systemic vasodilation which precipitates hepatorenal syndrome. Since systemic vasodilation plays a role in the development of ascites, bacterial byproducts via circulatory alterations may contribute to mechanisms leading to ascites formation. It is important to note that a randomized, double-blind, placebo-controlled trial of oral administration of the quinolone ciprofloxacin (500 mg/day for 1 year) has been conducted in a small series of patients with moderately severe cirrhosis, low ascitic fluid protein concentrations (<1.5 g/dL) and no prior history of SBP. However, ciprofloxacin therapy did not significantly increase the 1-year probability of being free of SBP. Taken together the findings of these 2 previous small-size trials suggest that long-term oral quinolone therapy is effective mainly in patients with severe cirrhosis. This is why we decided to perform a large multicenter, randomized, parallel, placebo-controlled trial assessing the effects of norfloxacin on survival in patients with cirrhosis and severe liver failure (Child-Pugh grade C). In addition, the effects of norfloxacin on the development of main complications of cirrhosis will be investigated.

The primary outcome measure will be 6-month survival. The secondary outcome measures will be the proportion of transplanted patients, the occurrence of complications (bacterial infection, renal failure, hepatic encephalopathy and gastrointestinal bleeding). All adult patients with severe cirrhosis might be randomized after written consent. Pregnant persons; patient who has been treated with a quinolone in the month before the inclusion, allergy to quinolones, hepatocellular carcinoma, or HIV infection will not be included. Patients receive either norfloxacin or placebo once a day for 6 months. Three hundred and ninety-two patients are necessary to decrease 6-month mortality rate from 40% in the placebo group to 25% in the norfloxacin group with a beta risk of 90% and an alpha risk of 5%. Patients will be followed-up every month during 6 months and at 9 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years,
* Liver failure as defined by a Child-Pugh score ≥ 10 points,
* Accept to participate,
* Have health insurance.

Exclusion Criteria:

* Pregnancy,
* Patient who has been treated with a quinolone in the month before his inclusion
* Allergy to quinolones,
* Hepatocellular carcinoma, and
* HIV infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 291 (Actual)
Dates: Start 2010-04; Primary Completion 2014-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Survival rate | 6 months

SECONDARY OUTCOMES:
Survival rate | 12-month follow-up
Number of patient with liver transplantation | 12 months
Complications : bacterial infection, renal insufficiency, hepatic encephalopathy, gastrointestinal bleeding | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: MOREAU RICHARD, Principal Investigator — APHP
Locations (1):
- Assisatnce publique Hoptitaux de Paris, Clichy, France

REFERENCES:
- [Derived] Moreau R, Elkrief L, Bureau C, Perarnau JM, Thevenot T, Saliba F, Louvet A, Nahon P, Lannes A, Anty R, Hillaire S, Pasquet B, Ozenne V, Rudler M, Ollivier-Hourmand I, Robic MA, d'Alteroche L, Di Martino V, Ripault MP, Pauwels A, Grange JD, Carbonell N, Bronowicki JP, Payance A, Rautou PE, Valla D, Gault N, Lebrec D; NORFLOCIR Trial Investigators. Effects of Long-term Norfloxacin Therapy in Patients With Advanced Cirrhosis. Gastroenterology. 2018 Dec;155(6):1816-1827.e9. doi: 10.1053/j.gastro.2018.08.026. Epub 2018 Aug 23. PMID 30144431